CLINICAL TRIAL: NCT07094152
Title: Blood Pressure Monitor (BPM1) Clinical Test (Cuff Range: 15cm-24cm, 22cm-42cm, 40-48cm)
Status: Completed | Type: Observational
Sponsor: Andon Health Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: Andon Health 15
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subject use both BPM1 Blood Pressure Monitor and mercury sphygmomanometers

SUMMARY:
The purpose of this study is to verify the accuracy of the blood pressure cuffs with blood pressure monitor device. Cuff circumference is: 15-24cm, 22-42cm, 40-48cm

ELIGIBILITY:
Inclusion Criteria:

* Normal blood pressure and hypertensive patients over 12 years old

Exclusion Criteria:

* Patients with serious arrhythmias or a high frequency of arrhythmias
* Pregnant woman
* Other investigators believe that it is not suitable to participate in this clinical trial

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Normal blood pressure and hypertensive patients over 12 years old
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2023-10-08 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Blood Pressure Monitor Accuracy | 30 minutes
  All the test results of the electronic blood pressure monitor with three (3) kinds of cuffs is within the accuracy creteria, with the merury sphygmomanometer as control

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, the Air Force Medical University, Xi’an, Shanxi, China